CLINICAL TRIAL: NCT07402525
Title: Postoperative Radiotherapy for Early-stage Oral Tongue Squamous Cell Carcinoma Patients With Risk Factors: a Prospective, Multicenter, Randomized Controlled, Open-labelled Trial
Acronym: PORT-ESTER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hunan Province Tumor Hospital (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sun Yat-sen University Cancer Hosptial (Unknown); Shanghai Cancer Hospital, China (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Xiangya Hospital of Central South University (Other); Sichuan Cancer Hospital and Research Institute (Other); Hunan Provincial People's Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The First Hospital of Jilin University (Other); First Hospital of China Medical University (Other); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Renmin Hospital of Wuhan University (Other); First Affiliated Hospital of Fujian Medical University (Other); Jiangxi Provincial Cancer Hospital (Other); Fujian Cancer Hospital (Other Government); Zhejiang Cancer Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Huzhou Center Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Huashan Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); The Second Affiliated Hospital of Harbin Medical University (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Qichun Wei, MD, PhD, professor of medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0846
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Oral Tongue Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PORT group (Experimental): Patients should start radiotherapy immediately after the surgical wound has fully healed, usually 4 to 6 weeks after surgery, with a requirement of no later than 8 weeks after surgery
  Interventions: Radiation: Postoperative radiotherapy
- control group (No Intervention): Patients will not receive special treatment and will undergo routine follow-up.

INTERVENTIONS:
Radiation: Postoperative radiotherapy — Radiation therapy should commence immediately after the surgical wound has fully healed, typically 4 to 6 weeks post-operation, but no later than 8 weeks post-operation
  Arms: PORT group

SUMMARY:
The goal of this clinical trial is to learn whether postoperative radiotherapy can delay disease recurrence in patients with early-stage oral squamous cell carcinoma who have high-risk factors. The main question it aims to answer is: Is the clinical outcome of early-stage tongue squamous cell carcinoma patients with risk factors after tumor enlargement resection receiving postoperative radiotherapy better than that of patients with simple follow-up observation? How is the safety? Researchers will compare the postoperative radiotherapy group and the simple follow-up observation group to see if there are differences between the two groups in terms of 3-year disease-free survival rate, 5-year disease-free survival rate, overall survival rate, toxicity events, and quality of life.

Participants of postoperative radiotherapy group will receive postoperative radiotherapy 6-8 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 70 years old, gender not limited;
2. Newly treated patients (who have not undergone radiotherapy, chemotherapy, or targeted therapy before);
3. Complete resection of the tumor with naked eye and no residual tumor observed in postoperative pathology;
4. The lesion is limited to the anterior 2/3 of the tongue (active part of the tongue);
5. Postoperative pathological diagnosis was squamous cell carcinoma of the tongue;
6. According to AJCC 8th edition, the pathological TNM staging is T1-2N0M0;
7. Having at least one risk factor: vascular cancer thrombus, nerve invasion, moderate or low differentiation;
8. The general status score of the Eastern Cancer Collaboration Group (ECOG) is 0-2 points;
9. Not participating in other clinical trials within the previous 4 weeks prior to screening; If other trials fail to screen cases, but meet the requirements of this trial, they can be enrolled.

Exclusion Criteria:

1. Patients who invade the oropharynx, mouth floor, cheeks, neck, and other organs;
2. Have received chemotherapy or other anti-tumor drugs;
3. Previously received radiation therapy for the head and neck area;
4. Patients with active autoimmune diseases that require systemic treatment in the past;
5. Pregnant or lactating women;
6. Individuals with acute infections that are difficult to control;
7. Patients with drug abuse, drug abuse, long-term alcoholism and AIDS;
8. The subjects also have other known invasive malignant tumors (excluding those with no evidence of tumor recurrence through treatment and a duration of more than 2 years);
9. Researchers believe that there are other conditions that hinder patients from participating in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2031-01-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
3-year DFS | 3 years
  The survival time of patients without significant tumor growth from the date of randomization. The appearance of new lesions is used as the criterion for recurrence (including recurrence of the primary lesion and surrounding tissues, cervical lymph node metastasis, and distant metastasis), and the time point of recurrence is the date of the first observation of measurable new lesions. The disease-free survival period will be defined as the time from randomization to death for patients who die from any other cause before disease recurrence is recorded. Patients who have not experienced disease recurrence or death (i.e. disease-free survival) during analysis will have the time of the last efficacy evaluation as the endpoint. For disease-free survival patients who have not undergone tumor evaluation since the baseline period, the first day of treatment will be used as the endpoint of disease-free survival. Calculate the 3-year disease-free survival rate of all patients after follow-up.

SECONDARY OUTCOMES:
5-year OS | 5 years
  From the date of randomization to the time of death caused by any reason. When recording lost patients until death, up to the last recorded time of contact with the patient. For patients who are still alive at the final analysis time point, their last contact time will be used as the survival time. During the analysis of survival and subsequent treatment, all patients were followed up until death, loss to follow-up, or termination of the study. The log rank test will be used to analyze the 5-year overall survival of all participants.
5-year DFS | 5 years
  The definition is the same as above. Calculate the 5-year disease-free survival rate of all patients after follow-up.
acute toxicity events | 6 months
  Evaluate toxicity events within 6 months after radiotherapy according to the RTOG acute radiation injury grading criteria and CTCAE v5.0 criteria.
Long-term toxicity events | from 6 months after treatment to 5 years after treatment
  according to CTCAE 5.0
scores of Quality of life | From enrollment to 5 years
  according to The University of Washington Quality of Life 4.0

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Chaoyang, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Cancer prevention and treatment center, sun yat-sen university, Guandong, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan cancer hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - The Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital & Institute, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The first affiliated hospital, college of medicinle, Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - the second affiliated hospital of Zhejiang University Hangzhou, Zhejiang, China, 310009, Hangzhou, Zhejiang
  - Huzhou Center Hospital, Huzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Xiangya Hospital of Central South University, Changsha
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou

IPD SHARING:
Plan to Share IPD: Undecided